CLINICAL TRIAL: NCT03337269
Title: Effectiveness of Targeted Educational Interventions at Increasing HPV Vaccine Acceptability and Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 826486
Record Dates: First submitted 2017-09-13; First posted 2017-11-08 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: HPV-Related Cervical Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Subject does not receive an educational intervention
  Interventions: Other: Control
- Educational video (Other): Subject watches an educational video
  Interventions: Other: Educational video
- Educational handout (Other): Subject reads an educational handout
  Interventions: Other: Educational handout

INTERVENTIONS:
Other: Educational video — Approximately 7 minute video on the HPV vaccine
  Arms: Educational video
Other: Educational handout — One page handout on the HPV vaccine
  Arms: Educational handout
Other: Control — Control
  Arms: Control

SUMMARY:
This study aims to assess the effectiveness of targeted educational interventions in increasing the acceptability and knowledge of the HPV vaccine among females ages 12 through 26. Subjects will be randomized to one of three study arms (no intervention, viewing an educational video or reading an educational handout) and then a questionnaire will be administered to assess knowledge and acceptability of the HPV vaccine. Subject charts will be reviewed to assess for initiation of the HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Females ages greater than or equal to 12 years and less than or equal to 26 years
2. Presenting to a gynecology clinic for a routine or problem visit
3. Ability to read and write

Exclusion Criteria:

1. Women ages less than or greater than 12 years or greater than 26 years
2. Women with known cervical cancer
3. Known pregnancy
4. Prior initiation or completion of the HPV vaccine series

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 256 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
HPV vaccine acceptability | Up to 6 months
  Subject reported willingness to accept the HPV vaccination, as assessed through agreement or disagreement to the statement "I would be willing to accept the HPV vaccine today."

SECONDARY OUTCOMES:
HPV vaccine knowledge | Up to 6 months
  Subject knowledge of the HPV vaccine and its associated risks and benefits, as assessed through a survey. Subjects are asked to answer 7 questions and total knowledge score is calculated by an unweighted sum of correct answers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cory L, Cha B, Ellenberg S, Bogner HR, Hwang WT, Smith JS, Haggerty A, Morgan M, Burger R, Chu C, Ko EM. Effects of Educational Interventions on Human Papillomavirus Vaccine Acceptability: A Randomized Controlled Trial. Obstet Gynecol. 2019 Aug;134(2):376-384. doi: 10.1097/AOG.0000000000003379. PMID 31306313